CLINICAL TRIAL: NCT02646787
Title: Water Friendly Virtual Reality for Burns
Brief Title: Virtual Reality Water Friendly Wound Care
Acronym: H2OWC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); University of Texas (Other)
Responsible Party: Principal Investigator, David Patterson, Professor, School of Medicine, Rehabilitation Medicine:Psychology, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002594; R01GM042725 (NIH)
Record Dates: First submitted 2015-12-15; First posted 2016-01-06 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Exergaming

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Virtual Reality (Experimental): The subject is actively engaged in using virtual reality during a painful burn wound care session.
  Interventions: Behavioral: Active Virtual Reality
- Passive Virtual Reality (Experimental): The subject is passively engaged in using virtual reality during a painful burn wound care session.
  Interventions: Behavioral: Passive Virtual Reality
- Control (No Intervention): No intervention during the subject's standard wound care session

INTERVENTIONS:
Behavioral: Active Virtual Reality — The subject is actively engaged in using virtual reality during a painful burn wound care session.
  Arms: Active Virtual Reality
Behavioral: Passive Virtual Reality — The subject is passively engaged in using virtual reality during a painful burn wound care session.
  Arms: Passive Virtual Reality

SUMMARY:
Using virtual reality as a form of distraction during a painful burn wound care procedure in addition to pain medication.

DETAILED DESCRIPTION:
Using virtual reality as a form of distraction during a painful burn wound care procedure in addition to pain medication.The aim of this study is to conduct a randomized controlled trial of Virtual Reality as a means to reduce pain during wound care in patients hospitalized for their burn injuries at Harborview Medical Center Burn Center, and Shriners Hospitals for Children in Galveston, Texas.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 8 years
* Compliant and able to complete questionnaires
* No history of psychiatric disorder
* Not demonstrating delirium, psychosis or any form of Organic Brain Disorder
* Able to communicate verbally
* English-speaking

Exclusion Criteria:

* Age less than 8 years
* Not capable of indicating pain intensity
* Not capable of filling out study measures
* Evidence of traumatic brain injury
* History of psychiatric disorder
* Demonstrating delirium, psychosis or any form of Organic Brain Disorder and associated memory problems
* Unable to communicate orally
* Receiving prophylaxis for alcohol or drug withdrawal
* Developmental disability
* Any face/head/neck injuries that interfere with the use of Virtual Reality equipment
* Non-English Speaking
* Extreme susceptibility to motion sickness
* Seizure history

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Pain. Pain is measured one time prior a painful burn wound care session, by asking the subjects about their pain level, using a questionnaire called graphic rating scale. | one time for the duration of one minute before the wound care
Pain. Pain is measured one time after a painful burn wound, by asking the subjects about their pain level, using a questionnaire called graphic rating scale. | one time for the duration of one minute after the wound care

CONTACTS AND LOCATIONS:
Overall Officials: David R Patterson, Ph.D., Principal Investigator — University of Washington; David R Patterson, Ph. D., Principal Investigator — University of Washington
Locations (1):
- University of Washington; Harborview Medical Center, Seattle, Washington, United States